CLINICAL TRIAL: NCT05384327
Title: Development and Validation of a Theoretical Test for Chest Tube Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ID 5046
Record Dates: First submitted 2022-05-13; First posted 2022-05-20 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Chest Tubes; Cognitive Skill
Keywords: Chest Tube; Assessment
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Interview (Other): Content experts who will be interviewed in order to collect their opinion on theoretical knowledge.
  Interventions: Other: Interview
- Novices (Other): Medical students who will complete the test
  Interventions: Other: Multiple Choice Question (MCQ) Test
- Intermediates (Other): Junior residents (surgery, pneumology, emergency medicine) who will complete the test.
  Interventions: Other: Multiple Choice Question (MCQ) Test
- Experienced (Other): Faculty members (surgery, pneumology, emergency medicine) who will complete the test.
  Interventions: Other: Multiple Choice Question (MCQ) Test

INTERVENTIONS:
Other: Interview — Interviews consist of semi-structured interviews focused on the theoretical knowledge a physician should possess before placing chest tube insertions.
  Arms: Interview
Other: Multiple Choice Question (MCQ) Test — The test contains multiple choice questions based on these interviews. Participants will complete this test.
  Validity evidence will be collected based on the results of this test.
  Arms: Experienced; Intermediates; Novices

SUMMARY:
The goal of the proposed study design is to develop and gather validity evidence of a theoretical test about cognitive skills which are important when performing Chest Tube Insertion (CTI). This study consists of two parts:

* The development of the theoretical test and its items. The test content will be based on a broad literature search, and on semi-structured interviews with content experts.
* The subsequent collection of validity evidence for this theoretical test and final selection of the test items, by testing groups that differ based on their expertise. The item analysis and observed difference in mean score between the groups will provide the validity evidence.

ELIGIBILITY:
Inclusion Criteria:

* Content experts will be recruited from the departments of surgery, pulmonology, and emergency medicine of various hospitals in Flanders and the Netherlands. They must have finished their residency training and be actively involved in training of junior physicians. A maximum of six experts will be recruited, and a minimum of one physician from each department will be included.
* The novice group will attract medical students at Ghent University, within their 5th or 6th year of undergraduate training, while having no experience with CTI.
* The intermediate group will include residents of the departments of surgery, pulmonology and emergency medicine of Ghent University Hospital, within their 1st - 3rd year of residency training and must have placed less than 20 chest tubes themselves.
* The experienced group will be recruited from the departments of surgery, pulmonology, and emergency medicine of Ghent University Hospital. They must have finished the residency training in their respective fields and must have performed more than 20 CTI independently. The content experts will not be eligible for participation.

Exclusion Criteria:

* For the novice and intermediate group: having to much experience in CTI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Validity evidence for the theoretical test | Participants are assessed once: the score of each participant is recorded immediately after completion of the test.
  Validity evidence following Messick's framework for a new theoretical test will be collected. The score will reflect the number of questions participants scored correctly; X/Y, where X=the number of questions answered correctly, and Y=the total number of questions. This score can be transformed in a percentage score accordingly. A higher score means the participant answered more questions correctly.

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Willaert, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No